CLINICAL TRIAL: NCT01344096
Title: A 1.5 Years Prospective Study Designed to Delineate the Cause of the Thrombocytopathy in Gaucher Disease Patients
Brief Title: Thrombocytopathy in Gaucher Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: RMC6088; GZGD02507 (Other Grant/Funding Number: Genzyme)
Record Dates: First submitted 2011-03-14; First posted 2011-04-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Gaucher Disease; Thrombocytopathy
Keywords: Gaucher disease; Thrombocytopathy; Imiglucerase
MeSH Terms: conditions — Gaucher Disease; Blood Platelet Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
In Gaucher disease type I bleeding is a common presenting symptom, that may manifest itself as frequent nose bleeds, easy bruising but can also cause substantial bleeding after surgical or dental procedures and may occur in association with pregnancy or delivery . The bleeding tendency is usually considered to be secondary to thrombocytopenia However 50,000 platelets are enough in healthy people to give a normal bleeding time but are associated with significant bleeding tendencies in Gaucher patients. Bleeding tendency might be attributed by genetic inherited or Gaucher related coagulation factors abnormalities which in some cases stabilize with ERT. However, In other cases the etiology is an abnormality of platelet function. This thrombocytopathy has not been delineated and apart from a few aggregation studies, no systematic analysis has been published that convincingly shows the cause of the disturbed function. While, experience shows that enzyme replacement (ERT, i.e: imiglucerase, Cerezyme®) reduces this bleeding tendency, in part due to the improvement in the thrombocyte count and elevation in coagulation factors, it is less clear what effect ERT has on the thrombocytopathy. This has clinical significance when patients need to be prepared for surgery or delivery or in the event of a major bleed. There is no consensus as to how patients should be prepared or treated. Different centres use different approaches. When the procedure is elective ERT is appropriate but in other situations DDAVP, fresh frozen plasma and platelet infusion are possible treatments. Even activated factor VII has been used when bleeding was not controlled. As in any other coagulation abnormality, treatment should be tailored to the specific cause of the bleeding diathesis. The aim of this study is to define the etiology of platelet dysfunction in Gaucher patients.

Hypothesis: The investigators expect to see a difference between platelets activation profile among imiglucerase treated and untreated patients with at least a partial restoration of platelets function due to treatment commencement.

DETAILED DESCRIPTION:
Objectives:

Delineating the cause of the thrombocytopathy in Gaucher disease patients:

1. Identifying thrombocytopathy among a cohort of 70 Gaucher patients managed (treated and untreated) in our clinic using a panel of platelets function tests.
2. Understanding the etiology for platelets dysfunction in Gaucher disease.
3. Evaluating the impact of Imiglucerase treatment duration and Gaucher disease severity on platelet function

ELIGIBILITY:
Inclusion Criteria:

* Gaucher disease patients
* Patients who do not receive any medicine that affects platlats

Exclusion Criteria:

* Treatment with enzyme replacement therapy other than Imiglucerase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gaucher disease patients treated and untreated wih Imiglucerase
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-10; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Measure thrombocytopathy in a cohort of 70 Gaucher patients using a set of platelet function tests. | 3 years
  • 70 Gaucher patients managed (treated and untreated controls) will be subjected to a panel of platelets function tests (aggregation test, closure time and FACS analysis).

SECONDARY OUTCOMES:
Evaluating the impact of Imiglucerase treatment on platelet function | 3 years
  Platelet function during the 3 years of study will be analyzed versus Imiglucerase treatment status and duration taking into consideration genotype, age at diagnosis, spleen status and Gaucher disease severity at treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Cohen, Prof., Study Chair — Rabin Medical Center; Hagit Baris, MD, Study Chair — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva

REFERENCES:
- [Derived] Baris HN, Weisz Hubshman M, Bar-Sever Z, Kornreich L, Shkalim Zemer V, Cohen IJ. Re-evaluation of bone pain in patients with type 1 Gaucher disease suggests that bone crises occur in small bones as well as long bones. Blood Cells Mol Dis. 2016 Sep;60:65-72. doi: 10.1016/j.bcmd.2015.05.003. Epub 2015 May 9. PMID 26051481